CLINICAL TRIAL: NCT01644357
Title: Effect of a 12-month Pharmaceutical Care Program on Severe Asthma Patient. A Randomized Clinical Trial
Brief Title: Effect of a 12-month Pharmaceutical Care Program on Control of Severe Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Pablo de Moura Santos, Pharmacist, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ATENFAR-PROAR
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Asthma; Quality of Life
MeSH Terms: conditions — Asthma | interventions — Pharmaceutical Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dispensing only (No Intervention): Non clinical pharmacists will dispense drugs to patients and usual care will be offered.
- Pharmaceutical care (Experimental): Patients on experimental group will receive counseling and education on the asthma condition, medication and lifestyle issues. In all visits, the inhaler technique will be reviewed, adherence to treatment and drug related problems were checked. If necessary the patient will be referred to the respiratory specialist to change the medication or to prescribe dose adjustment. Pharmacists document their initial and monthly follow up encounters using a specified form.
  Interventions: Other: Pharmaceutical care

INTERVENTIONS:
Other: Pharmaceutical care — Pharmacist intervention, focused on the optimization of drug therapy, identification and resolution of drug related problems, resulting in best asthma control and quality of life. Pharmacists document their initial and monthly follow up encounters using a specified form. An action plan for self management of these patients was prepared and discussed aiming at early identification and treatment of an exacerbation episode. Meetings will be held weekly with intervention team to discuss action plan and measure of outcomes of all problems identified.
  Arms: Pharmaceutical care

SUMMARY:
Only a few well-designed studies have investigated the effect of pharmaceutical care on asthma patients and to date there are no published studies investigating this effect specifically on severe and refractory asthma.

The objective of this study is evaluate the effect of pharmaceutical care on asthma control and quality of life (QoL) of patients with severe or refractory asthma compared with pharmacist dispensation only.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe/refractory asthma presenting other respiratory disease,
* ≥ 18 years of age,
* using high dose of inhaled corticosteroids (≥ 800mcg of budesonide or equivalent)
* FEV1<60%,
* regular visitor of the pharmacy and the physicians.

Exclusion Criteria:

* participation in other intervention study during this study,
* living in other cities,
* could not participate in all visits of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2011-08 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
asthma control of symptoms | 12 months
  Measured by Asthma Control Questionnaire and medical evaluation

OTHER OUTCOMES:
Lung function improvement | 12 months
  Measured by spirometry
Quality of life improvement | 12 months
  Measured by Asthma Quality of Life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pablo M Santos, Master, Principal Investigator — Federal University of Bahia; Álvaro A Cruz, Professor, Study Director — Federal University of Bahia; Lúcia B Noblat, Professor, Study Chair — Federal University of Bahia
Locations (1):
- Program for Asthma Control (ProAR) of the Federal University of Bahia, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No
Publish a paper in a cientific journal